CLINICAL TRIAL: NCT06464094
Title: User-Testing Protocol for the Cloud DX Vitaliti Continuous Vital Signs Monitor (Model CVSM-1A) for Clinical Use and Self Measurement in Ambulatory Settings
Brief Title: Vitaliti Continuous Vital Signs Monitor User-Testing Protocol: VERDICT-2
Acronym: VERDICT-2
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: McMaster University (Other); Population Health Research Institute (Other); Cloud DX Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 3.0_2023.05.31
Record Dates: First submitted 2024-06-05; First posted 2024-06-18 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Surgery
Keywords: User-testing; Device

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- User-testing of Vitaliti Continuous Vital Sign Monitor Model CVSM-1A (Other): Participants enrolled to engage in user-testing of the Vitaliti Continuous Vital Sign Monitor Model CVSM-1A to examine user-acceptance and user experiences, while soliciting user feedback on wearability compliance (patient) and proposed clinical workflows using the most recent Vitaliti™ CVSM device.
  Interventions: Other: User-testing of Vitaliti Continuous Vital Sign Monitor Model CVSM-1A

INTERVENTIONS:
Other: User-testing of Vitaliti Continuous Vital Sign Monitor Model CVSM-1A — Single group enrollment to examine user-acceptance and user experiences, while soliciting user feedback on wearability compliance (patient) and proposed clinical workflows using the most recent Vitaliti™ CVSM device.

SUMMARY:
The VERDICT-2 user testing study will user test the Cloud DX Vitaliti Continuous Vital Signs Monitor (Model: CVSM-1A) in an ambulatory context with post-surgical participants, their family members (caregiver support role) and clinicians (nurses and physicians) at Hamilton Health Sciences to examine user acceptance and user experiences, while soliciting user feedback on wearability compliance and proposed clinical workflows.

DETAILED DESCRIPTION:
Effective postoperative care is faced with several challenges- patients experience major complications following surgery, which often require re-hospitalization or utilization of healthcare services (i.e., emergency room visits) once discharged into the community. New remote automated monitoring (RAM) technologies that enable data integration, synthesis, and real-time alerts to clinicians have the potential to transform postoperative care, similar to how intraoperative care has evolved.

The Cloud DX Vitaliti Continuous Vital Signs Monitor (Model: CVSM-1A) is a continuous vital sign monitor intended to measure vital metrics including systolic and diastolic blood pressures (via ECG/ photoplethysmography [PPG]), pulse (via PPG), respiration rate (via impedance respiration waveform), core body temperature (via infrared sensor), and blood oxygen saturation levels (via PPG) of an adult individual using non-invasive techniques.

The VERDICT-2 user testing study will user test the Cloud DX Vitaliti Continuous Vital Signs Monitor (Model: CVSM-1A) in an ambulatory context with post-surgical participants, their family members (caregiver support role) and clinicians (nurses and physicians) at Hamilton Health Sciences to examine user acceptance and user experiences, while soliciting user feedback on wearability compliance and proposed clinical workflows.

ELIGIBILITY:
Patient Inclusion Criteria

1) Age ≥45 years; 2) Undergoing inpatient non-cardiac surgery with general or regional anesthesia; 3) Expected to spend at least two nights in hospital after surgery; 4) Provide written informed consent to participate in the VERDICT-2 Study, AND 5) Fulfill ≥ 1 of the following criteria (a-e):

a. History of coronary heart disease; b. History of stroke; c. History of peripheral arterial disease; d. Preoperative NT-proBNP value ≥200 ng/L e. OR fulfill ≥3 of the following 9 risk factors: i) Undergoing major surgery ii) Undergoing urgent or emergent surgery iii) History of hypertension iv) History of congestive heart failure v) History of transient ischemic attack vi) History of smoking within 2 years of surgery vii) Diabetes and currently taking an oral hypoglycemic agent or insulin viii) Age >70 years

Patient Exclusion Criteria

1. Intolerance/allergy to adhesive
2. Hearing aid/Cochlear Implant
3. Patients with cognitive or physical impairments hindering understanding the scope of the device or ability to interact with the device or unable to communicate with research staff, complete study surveys, or undertake an interview using technology will not be eligible for recruitment

Family/Care Giver Inclusion Criteria:

1. Age >18 years
2. Family or non-family member, residing in the same household as the patient or closely involved in the patient's postoperative recovery
3. Provide written informed consent to participate in the VERDICT-2 Study

Family/Care Giver Exclusion Criteria:

1) Caregivers with cognitive or physical impairments hindering understanding the scope of the device or ability to interact with the device or unable to communicate with research staff, complete study surveys, or undertake an interview using technology will not be eligible for recruitment

Clinician Inclusion Criteria:

1. Registered Nurse or Physician engaged in perioperative care
2. Employed at Hamilton Health Sciences
3. Provide written informed consent to participate in the VERDICT-2 Study

Clinician Exclusion Criteria:

1. Clinicians unable to understand the scope of the device or ability to interact with the device or unable to communicate with research staff, complete study surveys, or undertake an interview using technology due to language barriers will not be eligible for recruitment
2. Non-practicing class of licensure

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Task analysis | During user testing (Single sitting; 30-60 Minute duration)
  Assessment of all users' (patient, caregiver, clinician) performance of the required tasks during Vitaliti™ CVSM user testing according to the following designations: 'completed', 'completed with difficulty', or 'missed'. Descriptive data will be generated to summarize operational tasks that required the most support to complete.
Wearability (Patients) | 72 hours
  Participant journal used to record any device removal occurrences reason why it was taken off, and for how long. Participants will also be asked to keep track of any experiential information they note while wearing the device, which will then be provided to the research team for review.
Impressions of usability (Patients) | 72 hours (single sitting; 30-60 Minute interview)
  In-person post-test debrief interviews for patients, caregivers, and clinicians will be conducted using semi-structured interview methods following the task analysis user-testing exercise. These interviews will focus on perceptions of usability as they relate to root causes of sources of difficulty and particular events that may have occurred. Participants' overall impressions of the usability of the Vitaliti™ system will also be captured, focusing on perceived successes and failures, impressions of what may be done differently next time, as well as feedback on the in-service and training materials provided. Analysis by qualitative methods.
Impressions of usability (Caregivers) | 72 hour (single sitting; 30-60 Minute interview)
  In-person post-test debrief interviews for patients, caregivers, and clinicians will be conducted using semi-structured interview methods following the task analysis user-testing exercise. These interviews will focus on perceptions of usability as they relate to root causes of sources of difficulty and particular events that may have occurred. Participants' overall impressions of the usability of the Vitaliti™ system will also be captured, focusing on perceived successes and failures, impressions of what may be done differently next time, as well as feedback on the in-service and training materials provided. Analysis by qualitative methods.
Impressions of usability (Clinicians) | During user testing (single sitting; 30-60 Minute interview)
  In-person post-test debrief interviews for patients, caregivers, and clinicians will be conducted using semi-structured interview methods following the task analysis user-testing exercise. These interviews will focus on perceptions of usability as they relate to root causes of sources of difficulty and particular events that may have occurred. Participants' overall impressions of the usability of the Vitaliti™ system will also be captured, focusing on perceived successes and failures, impressions of what may be done differently next time, as well as feedback on the in-service and training materials provided. Analysis by qualitative methods.

CONTACTS AND LOCATIONS:
Locations (1):
- McMaster University, Hamilton, Ontario, Canada